CLINICAL TRIAL: NCT04393376
Title: Evaluation of Prostate-Specific Antigen Glycomics Assay for the Early Detection of Prostate Cancer
Brief Title: PSA Glycomics Assay for Early Detection of Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof.dr. H.P. Beerlage (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); The Netherlands Cancer Institute (Other); Radboud University Medical Center (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Prof.dr. H.P. Beerlage, Urologist, Head of Department of Urology, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL73261.018.20
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Prostate Cancer; PSA
Keywords: Prostate Cancer; PSA; Glycomics Assay
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PSA Glycomics Assay — PSA Glycomics Assay will be performed on urine and blood samples

SUMMARY:
The principal aim of this pilot study is to test whether the PSA Glycomics Assay on urine and serum samples can provide insights regarding the disease state of patients with elevated PSA concentrations, as well as to accurately identify if the patient has prostate cancer and, in the case of prostate cancer, to determine its level of aggressiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients with elevated PSA (>3 ng/mL)
* Signed informed consent

Exclusion Criteria:

* Patients that have a cystitis (bladder infection)
* Patients under chemotherapy
* Patients using 5-alpha reductase inhibitors
* History or presence of cancers, or non-prostate urological disorders.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
PSA Glycomics Assay | 1 year
  The relative abundance of glycoforms of PSA in plasma and urine from the subjects will be measured. These will be related to the stage of PCa and compared to non-prostate cancer patients.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Amsterdam UMC, location AMC, Amsterdam, North Holland
  - Amsterdam UMC, location VUmc, Amsterdam
  - Leiden University Medical Centre, Leiden

IPD SHARING:
Plan to Share IPD: Undecided